CLINICAL TRIAL: NCT05531123
Title: A Prospective Phase II Study of Risk-stratification Based Bladder-sparing Modalities for Muscle-invasive Bladder Cancer After Chemotherapy Combined With PD-1 Antibody(Rebirth)
Brief Title: Risk-stratification Based Bladder-sparing Modalities for Muscle-invasive Bladder Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, Professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ReBirth-01
Record Dates: First submitted 2022-08-29; First posted 2022-09-07 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — tislelizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1(cCR=cT0, cTa) (Experimental)
  Interventions: Drug: Tislelizumab
- Arm2 (non-cCR) (Experimental)
  Interventions: Drug: Tislelizumab; Drug: gemcitabine and cisplatin; Radiation: Modified hypofractionation

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200 mg I.V. Q3W on the day 1
Drug: gemcitabine and cisplatin — Cisplatin 70mg/m2 I.V. Q3W on the day 1, dose fractionation is allowed ;Gemcitabine 1000mg/m2 I.V. Q3W on the day 1 and day 8
  Arms: Arm2 (non-cCR)
Radiation: Modified hypofractionation — * Whole bladder 44Gy / 16fractionation (If N1: Whole bladder + Pelvic nodes 44Gy / 16fractionation) (Positive lymph nodes can be dosed to the maximum tolerable dose)
  * Tumor boost 11Gy / 4fractionation
  * Radiosensitizing chemotherapy: DDP 75-80 mg/m2 weekly Q3W
  Arms: Arm2 (non-cCR)

SUMMARY:
Neoadjuvant chemotherapy plus radical cystectomy is the standard if care for cisplatin-eligible patients with MIBC. Developments in the last two decades suggest that bladder sparing therapy may be a valuable alternative to radical cystectomy. Currently, well-documented TMT regimens, which include complete transurethral resection of bladder tumor (TURBT), chemotherapy, and radiation therapy, demonstrated durable oncologic control and long-term survival in selected patients. Nevertheless, TMT has not been widely used in clinical practice. On the one hand, due to the complexity of TMT, multiple clinical departments are required to cooperate in the assessment, treatment and follow-up of patients. On the other hand, concerns about tumor recurrence, lack of surgical intervention in regional lymph nodes, and organ dysfunction due to the treatment of large doses of pelvic radiation have reduced the clinical acceptance of TMT. In recent years, immunocheckpoint inhibitors such as PD-1/L1, including Nivolumab, Pembrolizumab, and Tislelizumab, have proven to be promising immunotherapy approaches for advanced urothelium cancer, leading to breakthroughs in the treatment of advanced urothelium cancer. Immunocheckpoint inhibitors also showed positive efficacy in patients who did not respond to BCG treatment during perioperative period. Therefore, immunotherapy can be another means of bladder preservation after surgery, chemotherapy and radiotherapy. However, bladder sparing target population is still unclear, among which, the NCCN guidelines recommend patients suitable for bladder preservation: T2-3N0M0, single lesion (longest diameter less than 6 cm), histological type of urothelial carcinoma, no CIS, and no hydronephrosis. Therefore, the focus of bladder preservation treatment is not only on the treatment before and during bladder preservation, but also on maximizing the follow-up treatment of TURBT and exploring its long-term benefits based on response to systematic treatment before maximized TURBT.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and ≤ 85;
* People who want to protect their bladder;
* ECOG PS 0 2 points;
* Subject underwent TURBT surgery and imaging diagnosis of musculothelial invasive bladder urothelial carcinoma (histologic variation accepted, not diffuse CIS lesion);
* Accept maximum TURBT;
* Clinical stages T2-4A, N0-1, M0;
* Normal function of major organs (14 days prior to enrollment), i.e. meeting the following criteria:

  1. Blood routine examination criteria should be met (no blood transfusion and no granulocyte colony were received within 14 days before enrollment Stimulator therapy) :

     HB 90 g/L or higher The ANC acuity 1.5 x 109 / L PLT acuity 100 x 109 / L
  2. No functional organic disease, the following criteria should be met:

T-bil ≤1.5×ULN upper limit of normal value ALT and AST≤2.5×ULN If liver metastasis, ALT and AST≤5×ULN Estimated glomerular filtration rate (EGFR 60mL /min MdRD formula) International standardized ratio (INR), activated partial thrombin time aPTT ≤1.5× ULN(this standard is only applicable to patients who did not receive anticoagulant therapy; On anticoagulant therapy Patients should keep anticoagulants within the therapeutic range)

* Men who are fertile or women who are likely to become pregnant must use highly fertile men or women who are likely to become pregnant during the trial, Must be used in the testing process highly effective contraceptive methods (such as oral contraceptives, intrauterine contraceptive device, abstemious sexual desire or barrier contraception effective contraceptive methods (such as oral contraceptives, intrauterine contraceptive device, abstemious sexual desire or barrier contraceptive method combined with spermicide), and at the end of the treatment to birth control in combination with spermicide), and birth control for 12 months after the end of the treatment;
* Subjects voluntarily joined the study and signed informed consent with good compliance and follow-up. The subjects voluntarily joined the study and signed informed consent with good compliance and follow-up.

Exclusion Criteria:

* Previously received anti-PD-1, anti-PD-L1, and anti-PD-L2 therapy;
* Known to be allergic to recombinant humanized anti-PD-1 monoclonal antibody drugs and their components;
* Received other antineoplastic therapy (including but not limited to corticosteroids) within 4 weeks prior to study therapy;
* Alcohol therapy, immunotherapy) or other clinical studies, or have not yet recovered from the previous toxicity (except 2 degree hair loss and 1 degree neurotoxicity);
* Women who are pregnant or breast-feeding, and women who wish to have children (pelvic radiation may cause ovarian function Premature aging);
* HIV positive;
* Patients with active hepatitis B or C; HBsAg or HBcAb positive patients were also detected with positive HBV DNA copy number (quantitative). The detection limit is 500IU/ml, or reaches the positive copy number detected by the research center); For such patients study screening must test for HBV DNA; HCV antibody test results are positive for patients, only when HCV RNA PCR test results. If it is negative, it can be included in this study;
* A clear history of active tuberculosis;
* Have active autoimmune diseases requiring systemic treatment within the past 2 years (e.g., using disease modulations);
* Section drugs, corticosteroids, or immunosuppressive drugs), allowing for relevant alternative therapies (e.g., thyroid Hormone, insulin, or physiological corticosteroid replacement therapy for renal or pituitary insufficiency);
* Other serious, uncontrolled comorbidities that may affect protocol compliance or interfere with interpretation of results;
* Diseases, including active opportunistic infections or advanced (severe) infections, uncontrolled diabetes, cardiovascular disease (Defined by the New York Heart Association classification as grade ⅲ or ⅳ heart failure, grade ⅱ or higher heart, visceral block, myocardial infarction in the past 6 months, unstable arrhythmia or instability, angina pectoris, cerebral infarction within 3 months, etc.) or lung diseases (interstitial pneumonia, obstructive pulmonary disease; History of pulmonary disease and symptomatic bronchial spasm);
* Received live vaccine within 4 weeks prior to the start of treatment;
* Prior allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
* Those who have a history of abuse of psychotropic substances and cannot quit or have a history of mental disorders; Those who have a history of psychotropic drug abuse and cannot quit or have a history of mental disorders;
* Large pleural or ascites with clinical symptoms or requiring symptomatic management; Large pleural or ascites with clinical symptoms or symptomatic management;
* In the past five years have suffered from other malignant tumors, not cured but does not include has obvious cured malignant swell years suffered from other malignant tumors, not cured but does not include has obvious cure of malignant tumor, or can cure cancer, such as basal skin cancer or squamous cell cancer, limitations before low-risk tumor, or can be a cure for cancer, Such as basal or squamous cell skin cancer, localized low-risk prostate cancer, cervical carcinoma in situ or breast carcinoma in situ; Remarks: Localized low-risk prostate cancer (defined as adenocarcinoma, carcinoma in situ of the cervix, or carcinoma in situ of the breast; Remark: Limits (defined as low-risk prostate cancer stage for stage or less T2a, gleason score, gleason scores six points or less, and diagnosis of prostate cancer and prostate cancer diagnosis in the PSA 10 ng/mL or less (such as test (e.g., measurement) of the patients received radical amount) of the patients received radical surgery operation and without prostate specific antigen (and prostate specific antigen (P SA)) biochemical relapses biochemical relapses may participate in this study); Participants may participate in this study);
* Previous history of pelvic radiation therapy; Previous history of pelvic radiation therapy;
* Merged UTUC or urethral cancer
* May increase risks associated with study participation, or may interfere with study participation, according to the researchers. Any other serious, acute or chronic medical or mental illness or laboratory abnormality that may increase the risk associated with study participation or that may interfere with the interpretation of study results or the interpretation of laboratory findings.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-10 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
BIDFS at one year | one year
  BIDFS, bladder intact disease free survival, was defined as the time from the start of regimen until MIBC recurrence, regional pelvic recurrence, distant metastasis, bladder cancer-related death, or cystectomy.

SECONDARY OUTCOMES:
MFS at two years | two years
  MFS, metastatic free survival, was defined as time from the start of regimen to first diagnosis of distant metastasis
BIDFS at two years | two years
  BIDFS, bladder intact disease free survival, was defined as the time from the start of regimen until MIBC recurrence, regional pelvic recurrence, distant metastasis, bladder cancer-related death, or cystectomy.
Treatment-related adverse events | two years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
cCR after first treatment stage | two years
  cCR, clinical complete response, defined as cT0, which is clarified as negative cystoscope, negative urine cytology and no disease evidence on imaging at the end of the first phase of treatment, and cTa, which is assessed as papillary bladder cancer by cystoscope, urine cytology and imaging.

OTHER OUTCOMES:
utDNA | two years
  Urine tumor DNA analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China